CLINICAL TRIAL: NCT04291664
Title: A Phase 1 PK and Dose Escalation and Expansion Study of DST-2970 in Patients With Prostate Cancer With Rising PSA on Treatment With Abiraterone Acetate
Brief Title: PK and Dose Escalation and Expansion Study of DST-2970
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dose escalation portion of the study completed, one expansion cohort was eliminated due to change in standard of care, and the second cohort was not enrolled based on future development considerations.
Sponsor: DisperSol Technologies, LLC (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DST-2970-104
Record Dates: First submitted 2019-11-27; First posted 2020-03-02 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; abiraterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prostate Cancer (Experimental)
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone 5Mg Tab; Drug: DST-2970 (Abiraterone)

INTERVENTIONS:
Drug: Abiraterone Acetate — Abiraterone Acetate 1000mg will be administered orally once daily
Drug: Prednisone 5Mg Tab — Prednisone 5mg will be administered orally twice daily with Abiraterone Acetate 1000mg
  Prednisone 5mg will be administered orally twice daily with DST-2970 for 28 days after dosing of Abiraterone Acetate is stopped
Drug: DST-2970 (Abiraterone) — DST-2970 will be administered orally twice daily for 28 days (for every cycle) after dosing of Abiraterone Acetate is stopped

SUMMARY:
This is a Phase I multi-center, open-label, study of DST-2970 to determine the MTD, overall safety/tolerability, PK/pharmacodynamic parameters, and efficacy in prostate cancer patients.The study will include a dose escalation phase followed by a dose expansion phase. Each cohort will consist of a "run-in" period to assess pharmacokinetic trough, as well as C1hour, C2hour, and C3hour levels of standard of care abiraterone acetate, followed by a minimum of an 80-hour washout (treatment delay), then initiation of treatment with DST-2970.

The patient population that will be evaluated in this study include patients with castration sensitive or castration resistant prostate cancer who experience a rising PSA, with or without radiographic progression, while taking abiraterone acetate.

In this protocol, "initial PSA response to abiraterone" is defined as having a ≥ 30% drop in PSA levels (confirmed by a second PSA level one month later) during the first 6 months of treatment with abiraterone. These patients who subsequently experience a rise in PSA while on abiraterone are considered as having "acquired resistance" to abiraterone in the context of this protocol. Patients not meeting the definition of having an "initial PSA response to abiraterone" are considered as having "primary resistance" to abiraterone in the context of the protocol.

In the dose escalation phase, all patients with a rising PSA can be enrolled, whether they had an "initial PSA response to abiraterone" or never responded to abiraterone.

Two expansion cohorts will be opened. One expansion cohort will evaluate patients who did achieve an "initial PSA response to abiraterone" within the first 6 months of treatment as defined above, but subsequently progressed by PSA with or without radiographic progression. A second expansion cohort will evaluate patients who did not achieve an "initial PSA response to abiraterone" as defined above but have PSA progression with or without radiographic progression.

The rationale of the study is to determine if the better bioavailability of DST-2970 will overcome resistance to abiraterone acetate experienced in these two clinical settings.

In all cohorts, treatment will continue until progressive disease, unacceptable toxicity, investigator and/or sponsor decision, intercurrent illness or patient withdrawal of consent.

Patients will be monitored regularly with physical examination and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients who have histologically or cytologically confirmed adenocarcinoma of the prostate (castrate sensitive or castrate resistant);

   1. During the dose escalation phase:

      Patients taking abiraterone acetate or enzalutamide as a single agent or in combination with Androgen Deprivation Therapy (ADT)
   2. During the expansion phase:

   Patients taking abiraterone acetate as a single agent or in combination with Androgen Deprivation Therapy (ADT).
2. Patients who have prostate-specific antigen (PSA) progression;

   1. During the dose escalation phase: Increasing PSA confirmed by 3 rising values (1.0 ng/mL minimum starting value) with or without radiographic progression
   2. During the dose expansion phase: Increasing PSA confirmed by sequence of rising values at a minimum of 1-week intervals (1.0 ng/mL minimum starting value) with or without radiographic progression
3. For the Expansion Cohorts

   1. Expansion Cohort 1: History of achieved an "initial PSA response to abiraterone" as defined in Section 3.1.
   2. Expansion Cohort 2: History of not having achieved an "initial PSA response to abiraterone as defined in Section 3.1.
4. Age ≥ 18 years.
5. ECOG Performance Status 0 or 1.
6. Patients must have the following laboratory values:
7. ANC > 1500/µL
8. Platelet count >100,000/µL
9. Hemoglobin > 9 g/dL
10. Bilirubin < 1.5 x upper limits of normal
11. ALT and AST < 2.5x upper limits of normal
12. Have acceptable renal function: calculated creatinine clearance ≥60 mL/min
13. Albumin > 2.8 g/dL.
14. Patient consent has been obtained according to local Institutional Review Board for acquisition of research specimens.
15. Patient is accessible and compliant for follow-up.
16. Patients with female partners of childbearing potential must agree to use barrier contraception (male condom) during the treatment period and for at least 30 days after the last dose.
17. Patient has a life expectancy of greater than 12 weeks.
18. Patient to be able to swallow the required tablets.

Exclusion Criteria:

1. For the Expansion Cohorts:

   1. Previous treatment with chemotherapy in the castrate resistant setting
   2. Positive for the ARV7 variant
2. History of failure after previous treatment with any androgen receptor blockers at any time (e.g., enzalutamide, apalutamide, darolutamide)

   a. Escalation Cohort: enzalutamide not excluded
3. Patients who had received previous therapy with ketoconazole for prostate cancer, lasting more than 7 days.
4. Have a corrected QT interval (using Fridericia's correction formula) (QTcF) of >450 msec in men
5. Have not recovered from adverse events (must be Grade ≤1) due to agents administered more than 4 weeks earlier.
6. Known hypersensitivity to any study drug component, or experienced grade 3 toxicity or higher with abiraterone acetate.
7. Concomitant use of strong CYP3A4 inducers unless these can be discontinued before enrollment into the study.
8. Concomitant use of sensitive CYP2D6 and CYP2C8 substrates unless these can be discontinued during the study (see Appendix 5)
9. Any concomitant condition that in the opinion of the investigator could compromise the objectives of this study and the patient's compliance.
10. Current malignancies of another type, with the exception of adequately treated in situ basal cell skin cancer or other malignancies with no evidence of disease for 2 years or more.
11. Known active HIV, HBV or HCV infection. Patients with a history of hepatitis B or C are allowed if HBV DNA or Hep C RNA are undetectable.
12. Documented or known serious bleeding disorder.
13. Clinically evident CNS metastases or leptomeningeal disease not controlled by prior surgery or radiotherapy; history of seizure disorder not controlled by anti-seizure medication at the time of enrollment. Patients with primary CNS malignancies are excluded.
14. Patients with a significant cardiovascular disease or condition, including:

    1. Myocardial infarction within 6 months of study entry
    2. NYHA Class III or IV heart failure, or known LVEF <50% (See Appendix 2)
    3. Uncontrolled dysrhythmias or poorly controlled angina.
    4. History of serious ventricular arrhythmia (VT or VF, ≥ 3 beats in a row) and/or risk factors (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
    5. Hypertension Grade 3 or higher. Patients with adequately treated hypertension are allowed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 26 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) | 12-18 Months
Recommended Phase II dose (RP2D) | 12-18 Months
Dose-Limiting Toxicity | 12-18 Months

SECONDARY OUTCOMES:
Pharmacokinetic analysis of trough, as well as C1hour, C2hour, and C3hour levels of abiraterone | 12-18 Months
  To evaluate the pharmacokinetic trough, as well as C1hour, C2hour, and C3hour levels of abiraterone following daily oral administration of DST-2970 to inform the dose selected for expansion in patients with prostate cancer
Change in Tumor Size | 12-18 Months
  To measure the effectiveness of DST-2970 using CT scan results as measured by modified RECIST 1.1
Change in Prostate Specific Antigen (PSA) | 12-18 Months
  To measure efficacy of DST-2970 using the blood marker PSA results
Duration of response (DoR) | 12-18 Months
  To measure duration of response (DoR)
Type of response (e.g., CR, PR, SD) | 12-18 Months
  To measure type of response (e.g., CR, PR, SD)
Time to Progression (rTTP) by PCWG3-modified RECIST v1.1 | 12-18 Months
  To measure Time to Progression (rTTP) by PCWG3-modified RECIST v1.1

OTHER OUTCOMES:
Exploration of potential biomarkers | 12-18 Months
  To explore potential biomarkers, including germline SNPs that may help predict response to DST-2970

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Miami, Miami, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Mays Cancer Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No